CLINICAL TRIAL: NCT05308056
Title: Depth of Anetshesia During Electroconvulsive Therapy
Brief Title: Depth of Anesthesia During Electroconvulsive Therapy
Acronym: ACDC
Status: Completed | Type: Observational
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: 276915
Record Dates: First submitted 2022-02-23; First posted 2022-04-01 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2022-02

CONDITIONS: Mood Disorders; Psychotic Disorders
Keywords: General anesthesia; Electroencephalogram; Awareness; Depth of anesthesia; Depression
MeSH Terms: conditions — Mood Disorders; Psychotic Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ECT-patients: Patients receiving routine ECT.
  Interventions: Device: Depth of anesthesia monitor, SedLine® (Masimo, Irvine, CA, USA)

INTERVENTIONS:
Device: Depth of anesthesia monitor, SedLine® (Masimo, Irvine, CA, USA) — The device monitors the patient's electroencephalogram using electrodes applied to the forehead.

SUMMARY:
Aim: To describe anesthetic depth using spectal edge frequency (SEF) and density spectral array (DSA) and its relation to treatment effect of electroconvulsive therapy (ECT).

Study design: Observational study Primary outcomes: SEF, DSA and treatment effect of ECT. Method: SEF and DSA si measured using a commercially available monitor for depth of anesthesia. Treatment effect of ECT will be evaluated using hemodynamic, electroencephalographic and clinical variables.

DETAILED DESCRIPTION:
Background Electroconvulsive therapy (ECT) is an effective therapy for severe depression where an electric current is applied to the brain to induce an epileptic seizure (1). The success of ECT is dependent upon the degree and quality of epileptic activity (2). ECT is normally administered after administering a muscle relaxant to prevent the seizure activity from causing muculoskeletal injuries. To tolerate the muscle relaxant the entire procedure is performed under general anesthesia. Most hypnotics have anti-convulsant effects and therefore counteract the effects of ECT (3). This implies that deep anesthesia hinders an optimal treatment effect of ECT which is supported by observational data (4). This relation has been proven with lighter anesthesia measured through bispectral index (BIS) correlating to longer seizure duration (5). BIS is not optimized to estimate the depth of anesthesia under very dynamic anesthetic protocols as there is an inherent latency in the computation of the BIS value. Anesthesia for ECT generally consists only of induction and recovery with no stable anesthetic phase making BIS an inappropriate measure of anesthetic depth. Indices of anesthetic depth that are derived directly from the processed EEG-signal have a negligent latency and can therefore be used with more precision during anesthesia for ECT. Spectral edge frequency (SEF) is the frequency under which 95 % of the total amplitude of the EEG-signal is found and it decreases with increasing depths of anesthesia. The density spectral array (DSA) is a graphic representation of the frequency and amplitude of the EEG signal over time and it is possible to interpret the DSA in real time without extensive training. The SEF and DSA have not, to our knowledge, been previously tested during general anesthesia for ECT. In the postictal phase during recovery from ECT some patients become agitated and confused (6). This condition is not clearly defined in the literature but is commonly referred to as postictal agitation (PIA) and due to differing definitions the incidence is difficult to estimate. Incidences in the range of 10-20 % have been reported (7). In the post-operative period after cardiac surgery decreased regional cerebral oxygen saturation (SrcO2) has been linked to post-operative confusion (8). A possible link between decreased SrcO2 and PIA has not been studied before.

Aim

The aim of this research project is two-fold:

1. To study the relation between anesthetic depth measured with SEF and DSA and the quality of epileptic activity during ECT.
2. To study the relation between SrcO2 and PIA during ECT.

Hypotheses

1. Lighter depths of anesthesia as measured by SEF and DSA have a positive correlation with epileptic seizure quality during ECT.
2. SrcO2 during ECT has an inverse correlation with the incidence of PIA. Method Setting and recruitment The study will be performed at the ECT-unit of the university hospital in Örebro. General anesthesia is provided by a nurse specially trained in anesthesia and an anesthesiologist. ECT is provided by specially trained nurses and staff at the ECT-unit. Patients recover from the postictal phase in an adjacent recovery room. Patients undergoing ECT through the outpatient clinic will be recruited to the study.

Anesthetic protocol The protocol for anesthesia and ECT will be the same as is being used clinically at the ECT-unit. After preoxygenation anesthesia is induced using thiopental. After confirmation of adequate anesthetic depth (failure to respond to verbal command) suxamethonium is administered. Doses are chosen by the anesthesiologist. Patients are admitted to the recovery room when breathing spontaneously and can maintain a patent airway.

Data collection SEF and DSA will be measured continuously from before pre-oxygenation to admittance to the recovery room using a SedLine® (Masimo, Irvine, CA, USA) monitor. The monitor will be blinded during the procedure so as not to affect the staff in any way. SrcO2 will be measured using the same monitor during the same period. Data regarding the seizure duration will be gathered from the electronic patient records. The staff caring for the postictal patients will estimate the degree of PIA according to previously used numerical scale (9).Data will be presented as mean ± SD or median (IQR) according to their distribution. Statistical analysis will be performed using a logistic regression model adjusted for potential confounders such as type of psychiatric medication, age, bilateral or unilateral stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for a course of ECT

Exclusion Criteria:

* Not able to attach electrodes for measurement of depth of anesthesia due to eg. skin condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted for ECT during the study period
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Change in spectral edge frequency | Monitored before, during and after ECT. Total monitoring time is apporximately 30 minutes per patient.
  The spectral edge frequency of the patients electroencephalogram
Change in density spectral array | Monitored before, during and after ECT. Total monitoring time is approximately 30 minutes per patient.
  The density spectral array of the patients electroencephalogram
Duration of convulsive activity | Monitored immediately after administration of ECT.
  Measures the duration of both motor and encephalographic convulsions directly following ECT.
Postictal supression | Monitored immediately after administration of ECT.
  Measures the degree of encephalographic supression directly following ECT
Need for restimulation | Monitored immediately after administration of ECT.
  Measures if there is a need for restimulation directly after evaluating the effect of an administered ECT.
Change in heart rate. | Monitored immediately after administration of ECT.
  Mesaures the increase in heart rate directly following ECT.

SECONDARY OUTCOMES:
Awareness | Patients are asked at a follow up visit approximately 1 week after a course of several ECT:s.
  Patients will be asked if they can recall any part of the tratment from induction of anesthesia until administration of ECT.
Adverse effects of ECT | Patients are asked at a follow up visit approximately 1 week after a course of several ECT:s.
  Occurence of adverse effects following ECT, evaluated using the CRPS-memory questionnaire.
Desaturation | Monitored immediately before pre-oxygenation, during the entire ECT and until the patient has recovered. Approximately 1 hours of total monitoring time.
  Occurence of saturation <92 % at any point during anesthesia and ECT.
End-tidal CO2 | During induction of general anesthesia
  Measurement of end-tidal CO2
Change in depressive symtoms | Patients are asked at a follow up visit approximately 1 week after a course of several ECT:s and before ECT.
  Effect of ECT on patients' symptoms and quality of life. Evaluated using the self-asessed Montgomery Åsberg Depression Rating Scale (MADRS-S), 0-57 points. A higher score indicate more severe disease.
Clinical assessment of depth of anesthesia | Monitored immediately before pre-oxygenation, during the entire ECT and until the patient leaves the recovery ward. Approximately 1 hour of total monitoring time.
  The treating anesthesiologist will be asked to asses the depth of anesthesia. The anesthesiologist is asked after induction of general anesthesia. The terms too heavily sedated, too lightly sedated and adequate level of sedation is used.
Regional cerebral oxygen saturation | Before, during and after anesthesia and ECT
  Measured using near-infrared spectroscopy
Occurence of post-ictal agitation | Monitored in the recovery suite
  Registered in the recovery ward following ECT. A scale using three levels of agitation is used by the recovery staff. Higher scores indicate increasing levels of agitation.
Change in quality of life | Patients are asked at a follow up visit approximately 1 week after a course of several ECT:s and before ECT.
  Effect of ECT on patients' symptoms and quality of life. Evaluated using EruroQol 5-Dimensions score (EQ-5D), each quiestion is scored 1-3 or 1-5 points. A higher score indicates worse health related problems.
Change in illness severity | Patients are asked at a follow up visit approximately 1 week after a course of several ECT:s and before ECT.
  Effect of ECT on patients' symptoms and quality of life. Evaluated using Clinial global impressions scale (CGI), each question is scored 1-7 points. A higher score indicates higher illness severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitetssjukhuset Örebro, Örebro, Bok 1613, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] UK ECT Review Group. Efficacy and safety of electroconvulsive therapy in depressive disorders: a systematic review and meta-analysis. Lancet. 2003 Mar 8;361(9360):799-808. doi: 10.1016/S0140-6736(03)12705-5. PMID 12642045
- [Background] Minelli A, Abate M, Zampieri E, Gainelli G, Trabucchi L, Segala M, Sartori R, Gennarelli M, Conca A, Bortolomasi M. Seizure Adequacy Markers and the Prediction of Electroconvulsive Therapy Response. J ECT. 2016 Jun;32(2):88-92. doi: 10.1097/YCT.0000000000000274. PMID 26397151
- [Background] Zolezzi M. Medication management during electroconvulsant therapy. Neuropsychiatr Dis Treat. 2016 Apr 19;12:931-9. doi: 10.2147/NDT.S100908. eCollection 2016. PMID 27143894
- [Background] Kronsell A, Nordenskjold A, Bell M, Amin R, Mittendorfer-Rutz E, Tiger M. The effect of anaesthetic dose on response and remission in electroconvulsive therapy for major depressive disorder: nationwide register-based cohort study. BJPsych Open. 2021 Mar 23;7(2):e71. doi: 10.1192/bjo.2021.31. PMID 33752777
- [Background] Guerrier G, Gianni MA. The effectiveness of BIS monitoring during electro-convulsive therapy: A systematic review and meta-analysis. J Clin Anesth. 2019 Dec;58:100-104. doi: 10.1016/j.jclinane.2019.05.006. Epub 2019 May 28. PMID 31151038
- [Background] Li X, Cheng N, Deng Y, Du J, Zhang M, Guo Y, Hei Z. Incidence and risk factors for postictal delirium in patients after electroconvulsive therapy in China. Asian J Psychiatr. 2020 Oct;53:102361. doi: 10.1016/j.ajp.2020.102361. Epub 2020 Aug 25. No abstract available. PMID 32890981
- [Background] Tsujii T, Uchida T, Suzuki T, Mimura M, Hirano J, Uchida H. Factors Associated With Delirium Following Electroconvulsive Therapy: A Systematic Review. J ECT. 2019 Dec;35(4):279-287. doi: 10.1097/YCT.0000000000000606. PMID 31764452
- [Background] Eertmans W, De Deyne C, Genbrugge C, Marcus B, Bouneb S, Beran M, Fret T, Gutermann H, Boer W, Vander Laenen M, Heylen R, Mesotten D, Vanelderen P, Jans F. Association between postoperative delirium and postoperative cerebral oxygen desaturation in older patients after cardiac surgery. Br J Anaesth. 2020 Feb;124(2):146-153. doi: 10.1016/j.bja.2019.09.042. Epub 2019 Dec 18. PMID 31862160